CLINICAL TRIAL: NCT00353457
Title: Phase II Study of Capecitabine, Oxaliplatin and Cetuximab Given Throughout Multi-Modal Therapy for Locally Advanced Rectal Adenocarcinoma
Brief Title: Capecitabine,Oxaliplatin & Erbitux Given Throughout Multi-Modal Therapy for Locally Advanced Rectal Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: new studies were finding that Erbitux was not beneficial
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 803437; UPCC 09204
Record Dates: First submitted 2006-07-14; First posted 2006-07-18 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Rectal Cancer
Keywords: Adjuvant therapy; Rectal cancer; Capecitabine; Oxaliplatin; Cetuximab; Erbitux
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Cetuximab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Capecitabine, Oxaliplatin and Cetuximab
  Interventions: Drug: Capecitabine, Oxaliplatin and Cetuximab; Radiation: Radiation

INTERVENTIONS:
Drug: Capecitabine, Oxaliplatin and Cetuximab — Capecitabine 825mg/m2 po BID D1-15 of 21 x2 cycles (Cyle 1 and 2), Capecitabine 825mg/m2 po BID weekly Sun PM-Fri AM x2 cycles (cycle 3 and 4), Capecitabine 825mg/m2 po BID D1-15 of 21 x4 cycles (cycle 5,6,7,8) Oxaliplatin 130mg/m2 IV Day 1 every 3 weeks x2 cycles (Cycle 1 and 2), Oxaliplatin 50mg/m2 IV weekly every Monday x2 cycles (Cycle 3 and 4), Oxaliplatin 130mg/m2 IV day 1 every 3 weeks x4 cycles (Cycles 5,6,7,8) Cetuximab 400mg/m2 IV cycle 1 day1, Cetuximab 250mg/m2 Day 1,8,15 of 21 for cycles 1-8
Radiation: Radiation — 45 Gy in 25 fractions, 3-fraction boost 5.4 Gy

SUMMARY:
This is a phase II study of induction chemotherapy (capecitabine, oxaliplatin and cetuximab (erbitux)) followed by capecitabine, oxaliplatin, cetuximab and radiotherapy followed by surgery followed by adjuvant capecitabine, oxaliplatin and cetuximab for locally advanced resectable rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed nonmetastatic, measurable, locally advanced (T3 or T4) rectal adenocarcinoma
* If available, tumor tissue must be sent for investigational immunohistochemical evaluations of EGFR status
* The distal border of the tumor must be at or below the peritoneal reflection (defined a with 12 cm of the anal verge by proctoscopy)
* Transmural penetration of the tumor demonstrated by CT + endorectal ultrasound or MRI
* ECOG PS 0-2
* No prior chemotherapy, biologic therapy or radiation therapy
* Age >= 18 years old
* Laboratory values: ANC >= 1500/mm3; Platelets >= 100,000/mm3; Hgb >= 9 g/dL; Estimated CrCl > 50 mL/min; Serum bilirubin <= 1.5 x ULN; AST and ALT <= 3.0 x ULN; Negative proteinuria based on dip stick reading
* Patients must either be not of child bearing potential or have a negative pregnancy test upon study enrollment. Patients must agree to continue contraception for 30 days from the date of the last study drug administration.

Exclusion Criteria:

* Pregnant or lactating woman. Women of childbearing potential with either a positive or no pregnancy test upon study enrollment. Women/men of childbearing potential not using a reliable and appropriate contraceptive method. Patients must agree to continue contraception for 30 days from the date of the last study administration.
* Life expectancy < 3 months
* Serious, uncontrolled, concurrent infection(s)
* Concurrent use of chemotherapy not indicated in the study protocol or any other investigational agents and patients who have received investigational drugs < 4 weeks prior to randomization.
* Prior therapy which specifically and directly targets the EGFR pathway.
* Prior severe infusion reaction to a monoclonal antibody
* Any prior therapy with Oxaliplatin
* Prior pelvic irradiation for any reason
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil or known DPD deficiency
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer
* Participation in any investigational drug study within 4 weeks preceding the start of the study treatment
* Major surgery within 4 weeks of the study treatment, without complete recovery
* Known, existing uncontrolled coagulopathy
* Unwillingness to give written informed consent
* Unwillingness to participate or inability to comply with the protocol for the duration of the study
* Known allergy or hypersensitivity to platinum-containing drugs
* Peripheral sensory neuropathy with functional impairment
* Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Pleural effusions or ascites that causes respiratory compromise
* Acute hepatitis or known HIV
* Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study: uncontrolled high blood pressure, history of labile hypertension, or history of poor compliance with anti-hypertensive regimen; unstable angina pectoris; symptomatic congestive heart failure; myocardial infarction < 6 months prior to randomization; serious uncontrolled cardiac arrhythmia; uncontrolled diabetes; active or uncontrolled infection; impairment of gastrointestinal function or GI disease that may significantly alter the absorption of Capecitabine.
* Evidence of CNS metastases or history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response | After neoadjuvant treatment

SECONDARY OUTCOMES:
Sphincter function | After surgery
Type of surgery | At time of surgery
Disease free survival | From time of study entry until first documented relapse

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Haller, M.D., Principal Investigator — Abramson Cancer Center of University of Pennsylvania; James M Metz, M.D., Principal Investigator — Abramson Cancer Center of University of Pennsylvania